CLINICAL TRIAL: NCT06018519
Title: A Prospective Study in Creatine Transporter Deficiency (SLC6A8) Patients to Determine the Most Relevant Outcome Measures
Brief Title: Relevant Outcome Measures for Creatine Transporter Deficiency Patient
Acronym: CREAT_criteria
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 69HCL21_0655; 2022-A02063-40 (Other: ID-RCB)
Record Dates: First submitted 2022-11-03; First posted 2023-08-30 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Creatine Transporter Defect
Keywords: Creatine Transporter Deficiency (SLC6A8); Outcome measures; Therapeutics; Feasibility; Relevance
MeSH Terms: conditions — Creatine deficiency, X-linked

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- CTD male patients (Other): Case group 24 male CTD patients having a confirmed mutation in the SLC6A8 gene, aged > 5 to < 35 years.
  Interventions: Other: Clinical endpoints; Other: Parental questionnaires; Other: Quality of life scale; Other: Cognitive assessments; Other: Language assessments; Other: Motor assessments; Other: Social assessments; Other: 3T MRI; Other: Cardiac assessments; Other: Biological collection
- Sex and chronological age matched male controls (Other): Control group 24 male, sex and chronological age matched controls, aged > 5 to < 35 years
  Interventions: Other: Clinical endpoints; Other: Cognitive assessments; Other: Language assessments; Other: Motor assessments; Other: Social assessments; Other: 3T MRI; Other: Biological collection
- Sex and mental age matched male controls (Other): Control group 24 male, sex and mental age matched controls, aged > 2 to < 8 years
  Interventions: Other: Clinical endpoints; Other: Cognitive assessments; Other: Language assessments; Other: Motor assessments; Other: Social assessments
- Typically developed children (Other): Control group 80 typically developed children aged > 2 to < 8 years, which corresponds to the mental age of CTD patients.
  40 children aged > 2 to < 5 years, and 40 children aged > 6 to < 8 years will perform the newly developed outcome measures.
  Interventions: Other: Cognitive assessments; Other: Language assessments; Other: Motor assessments; Other: Social assessments
- CTD female patients (Other): 15 female CTD patients having a confirmed mutation in the SLC6A8 gene, aged >5 to < 60 years
  Interventions: Other: Clinical endpoints; Other: Parental questionnaires; Other: Quality of life scale; Other: Cognitive assessments; Other: Language assessments; Other: Motor assessments; Other: Social assessments; Other: 3T MRI; Other: Cardiac assessments; Other: Biological collection
- Sex and mental age matched female controls (Other): Control group 15 female, sex and mental age matched controls, aged > 2 to < 8 years
  Interventions: Other: Clinical endpoints; Other: Cognitive assessments; Other: Language assessments; Other: Motor assessments; Other: Social assessments
- Sex and chronological age matched female controls (Other): Control group 15 female, sex and chronological age matched controls, aged > 5 to < 60 years
  Interventions: Other: Clinical endpoints; Other: Cognitive assessments; Other: Language assessments; Other: Motor assessments; Other: Social assessments; Other: 3T MRI; Other: Biological collection

INTERVENTIONS:
Other: Clinical endpoints — 1. Number of epileptic seizures
  2. Change in antiepileptic treatment (increase or decrease)
  3. Visual analogical scale on a target symptom defined with the parents,
  4. CGI,
  5. Actimetry data over 24 hours,
  6. Podometry data over 24 hours,
  7. 6 minutes' walk test,
  8. Clinical examination
  9. Feasibility of performing an MRI without any anesthesia on a mock scanner
  Arms: CTD female patients; CTD male patients; Sex and chronological age matched female controls; Sex and chronological age matched male controls; Sex and mental age matched female controls; Sex and mental age matched male controls
Other: Parental questionnaires — 10- Adaptive assessment with Vineland Adaptive Behavior scale II,
  11- Mac Arthur questionnaire regarding language,
  12- Pervasive Development Disorder in Mentally Retarded persons Scale (PDD-MRS),
  13- Dunn sensory profile,
  14- Aberrant Behavior Checklist,
  15- Nisonger Child Behavior Rating form,
  16- Social Responsiveness Scale 2,
  17- Scales assessing the impact on primary caregiver (CBI-M/ Beach Center Family QOL)
  Arms: CTD female patients; CTD male patients
Other: Quality of life scale — 18- Quality of life scale (PedsQL 4.0 for children or San Martin scale if the patient is older than 18)
  Arms: CTD female patients; CTD male patients
Other: Cognitive assessments — 19- Leiter 3 scale (4 cognitive sub-tests to be able to compute the non-verbal IQ and 2 non-verbal memory sub-tests) or Bayley 4 if Leiter 3 is not possible
  20- CPM-BF
  21- Simple reasoning task on tablet (match-to-sample task)
  22- Implicit rules learning (modified Brixton),
  23- 4 sub-tests from the WPPSI-IV ("zoo location" to assess spatial memory, "block design" to assess visuo-constructive abilities, "bug search" , "cancellation"),
  24- Attention assessment (4 sub-tests from KITTAP: alert, go/no go, flexibility, divided attention),
  25- Elementary visuo-spatial perception (on tablets)
Other: Language assessments — 26- EXALANG 3-6 (10 sub-tests testing for expressive and receptive language assessments),
  27- PPVT-5 (receptive vocabulary), EVT-3 (expressive vocabulary),
  28- Automatic language analysis (during a 10 minutes interaction, play).
Other: Motor assessments — 29- Kinematic task (specifically designed),
  30- Purdue-Pegboard test,
  31- Renzi test
Other: Social assessments — 32- Eye-tracking analysis of social visual scenes and social preference index (movies),
  33- theory of mind assessment,
  34- ADOS scale (Autism Spectrum Disorder),
  35- sensitivity to inequality,
  36- pro-social behaviors (help of the psychologist)
Other: 3T MRI — 37- Structural, metabolic and functional data
  Arms: CTD female patients; CTD male patients; Sex and chronological age matched female controls; Sex and chronological age matched male controls
Other: Cardiac assessments — 38- ECG
  39- Ultrasound
  Arms: CTD female patients; CTD male patients
Other: Biological collection — 40- Blood sample
  41- Urinary sample
  42- Superficial skin biopsy
  Arms: CTD female patients; CTD male patients; Sex and chronological age matched female controls; Sex and chronological age matched male controls

SUMMARY:
Creatine transport deficiency (CTD) is a rare genetic disorder related to pathogenic variants in the SLC6A8 gene, located on chromosome Xq28. Clinical diagnosis of CTD is based on clinical presentation, an increased urinary creatine/creatinine ratio and a severe decreased creatine peak on 1H-MRS magnetic resonance spectroscopy.

A retrospective study with questionnaires identified that most CTD patients had moderate to severe intellectual disability. Less than one third of patients were able to speak in sentences. Seizures were present in 59% of the patients. 41% had autistic features. Motor dysfunction was mentioned in 58%, and gastrointestinal symptoms were reported in 35% of the patients.

Several new therapeutic avenues are currently emerging in this disease for which no treatment has been available until now : cyclocreatine (interesting but unfortunately with very little clinical applicability due to its toxicity; dodecyl creatine ester incorporated into lipid nanocapsules with intranasal administration; pharmaco-chaperoning (for the folding-deficient creatine transporter variants, Ultragenyx pharmaceuticals new prodrug designed to deliver creatine to the brain (UX068). These new pharmacological treatment options may offer future opportunities to improve cognition in CTD patients.

A key issue is to determine outcome measures that are accessible to these patients, despite the importance of their cognitive deficit. In a preliminary study (on 31 CTD patients), investigators showed for example, that 75% of patients were unable to perform a Wechsler scale, which is one of the most used neuropsychological test to determine patient IQ (intelligence quotient). Most of the existing cognitive tests were developed to distinguish typically developing persons and ID (intellectual disability) patients, leading to a floor effect in the latter who systematically fail these tests. Therefore, these tests are not adapted to capture the potential effect of a drug in ID patient group. The identification of reliable and sensitive outcome measures for use in clinical trials in ID patients was recognized as a priority in a meeting convened by the NIH. N-of-1 trials (also called Single-Case Experimental Designs or SCEDs) appear of great interest for rare diseases, statistical power coming from the number of repeated measures, which leads to choose outcome measures that can be repeated multiple times.

This innovative study will allow to efficiently preparing future therapeutic trials, by specifying the phenotype of the patients, and by determining the most adapted outcome measures taking into account their cognitive deficiency and the type of experimental design to be used in the context of rare diseases.

ELIGIBILITY:
Inclusion Criteria:

Male CTD patients (n=24)

* Male CTD patients having a confirmed mutation in the SLC6A8 gene,
* Aged > 5 to < 35 years
* Whose maternal language is French,
* Having signed the informed consent and/or for whom parents/legal guardian have signed the informed consent,
* Affiliated to national Health Insurance system or parents/legal guardian affiliated to national health insurance system.

Female CTD patients (n=15)

* Female CTD patients having a confirmed mutation in the SLC6A8 gene,
* Aged > 5 to < 60 years,
* Whose maternal language is French,
* Having signed the informed consent and/or for whom parents/legal guardian have signed the informed consent.
* Affiliated to national Health Insurance system (sécurité sociale) or parents/legal guardian affiliated to national health insurance system

Sex- and chronological age-matched controls (n=24)

* Male
* Aged > 5 to < 35 years
* Whose maternal language is French,
* Having signed the informed consent and/or for whom parents/legal guardian have signed the informed consent,
* Affiliated to national health insurance system or parents/legal guardian affiliated to national health insurance system.

Sex- and chronological age-matched female controls (n=15)

* female,
* Aged > 5 to < 60 years,
* Whose maternal language is French,
* Having signed the informed consent and/or for whom parents/legal guardian have signed the informed consent
* Affiliated to national Health Insurance system (sécurité sociale) or parents/legal guardian affiliated to national health insurance system

Sex- and mental age-matched controls (n=39)

* Male and female
* Aged > 2 to < 8 years
* Whose maternal language is French,
* For whom parents/legal guardian have signed the informed consent,
* Affiliated to national health insurance system or parents/legal guardian affiliated to national health insurance system.

Typically developed children (n=80)

* Male and female
* Aged > 2 to < 8 years
* Whose maternal language is French,
* For whom parents/legal guardian have signed the informed consent,
* Affiliated to national health insurance system or parents/legal guardian affiliated to national health insurance system.

Sex- and chronological age-matched controls and Sex- and mental age-matched controls, aged < 8 years, could also be included in the Typically developed children group, as the data from the Typically developed children are only necessary to complete the developmental trajectory of the new tasks.

Non-inclusion Criteria:

CTD patients (n=39):

* Having a contraindication to the MRI examination (people using a pacemaker or an insulin pump, people wearing a metal prosthesis or an intracerebral clip, and claustrophobic subjects),
* Refusal of the subject and/or the subject's parents to be informed of possible abnormalities detected by MRI,
* Refusal of the subject and/or the subject's parents/legal guardian to be informed of possible abnormalities detected during the cardiac assessment.

Sex- and chronological age-matched controls (n=39)

* History of neurological or psychiatric disorder,
* Repetition of a grade,
* Learning disability requiring rehabilitation (speech therapy, psychomotor or oculomotor therapy),
* For participants agreeing on performing the MRI examination, having a contraindication to the MRI examination (use of a pacemaker or an insulin pump, people wearing a metal prosthesis or an intracerebral clip, and claustrophobic subjects) and refusal of the subject and/or the subject's parents/legal guardian to be informed of possible abnormalities detected by MRI.

Sex- and mental age-matched controls (n=39)

* History of neurological or psychiatric disorder,
* Repetition of a grade,
* Learning disability requiring rehabilitation (speech therapy, psychomotor or oculomotor therapy).

Typically developed children (n=80)

* History of neurological or psychiatric disorder,
* Repetition of a grade,
* Learning disability requiring rehabilitation (speech therapy, psychomotor or oculomotor therapy).

Ages: 2 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 197 (Estimated)
Dates: Start 2023-03-13 (Actual); Primary Completion 2026-12-13 (Estimated); Study Completion 2026-12-13 (Estimated)

PRIMARY OUTCOMES:
Clinical endpoints : number of epileptic seizures | Up to 90 Days
  Number of epileptic seizures
Clinical endpoints : antiepileptic treatment | For all 24 CTD patients: all examinations at V1 (Day 1/Day2) For 9 out of 24 CTD patients: examinations repeated every two weeks at V2 (Day15), V3 (Day30), V4 (Day45), V5 (Day60), V6 (Day75) and V7 (Day90).
  Change in antiepileptic treatment (increase or decrease)
Clinical endpoints : Visual analogical scale | Up to 90 Days
  Visual analogical scale on a target symptom defined with the parents,
Clinical endpoints : actimetry | Up to 90 Days
  Actimetry data over 48 hours
Clinical endpoints : podometry | Up to 90 Days
  Podometry data over 24 hours
Clinical endpoints : walk test | Up to 90 Days
  6 minutes' walk test
Clinical endpoints : Clinical examination | For all 24 CTD patients: all examinations at V1 (Day 1/Day2) For 9 out of 24 CTD patients: examinations repeated every two weeks at V2 (Day15), V3 (Day30), V4 (Day45), V5 (Day60), V6 (Day75) and V7 (Day90).
  Clinical examination
Clinical endpoints :Feasibility of performing an MRI | For all 24 CTD patients: all examinations at V1 (Day 1/Day2) For 9 out of 24 CTD patients: examinations repeated every two weeks at V2 (Day15), V3 (Day30), V4 (Day45), V5 (Day60), V6 (Day75) and V7 (Day90).
  Feasibility of performing an MRI without any anesthesia on a mock scanner
Parental questionnaires : Vineland Adaptive Behavior scale II | For all 24 CTD patients: V1 (Day1/Day2), For 9 out 24 CTD patients: repeated at V7 (Day90).
  Adaptive assessment with Vineland Adaptive Behavior scale II
Parental questionnaires : Mac Arthur questionnaire | For all 24 CTD patients: at V1 (Day1/Day2), For 9 out 24 CTD patients: repeated at V3 (Day30) and V7 (Day90).
  Mac Arthur questionnaire regarding language
Parental questionnaires : PDD-MRS | For all 24 CTD patients: at V1 (Day1/Day2), For 9 out 24 CTD patients: repeated at V7 (Day90).
  Pervasive Development Disorder in Mentally Retarded persons Scale (PDD-MRS)
Parental questionnaires : Dunn sensory profile | For all 24 CTD patients: at V1 (Day1/Day2), For 9 out 24 CTD patients: repeated at V3 (Day30) and V7 (Day90).
  Dunn sensory profile
Parental questionnaires : Aberrant Behavior Checklist | For all 24 CTD patients: at V1 (Day1/Day2), For 9 out 24 CTD patients: repeated at V2 (Day15), V3 (Day30), V4 (Day45), V5 (Day60), V6 (Day75) and V7 (Day90).
  Aberrant Behavior Checklist
Parental questionnaires : Nisonger Child Behavior Rating form | For all 24 CTD patients: at V1 (Day1/Day2), For 9 out 24 CTD patients: repeated at V7 (Day90).
  Nisonger Child Behavior Rating form
Parental questionnaires : Social Responsiveness Scale 2 | For all 24 CTD patients: at V1 (Day1/Day2), For 9 out 24 CTD patients: repeated at V7 (Day90).
  Social Responsiveness Scale 2
Parental questionnaires : impact on primary caregiver | For all 24 CTD patients: at V1 (Day1/Day2), For 9 out 24 CTD patients: repeated at V3 (Day30) and V7 (Day90).
  Scales assessing the impact on primary caregiver (CBI-M/ Beach Center Family QOL)
Quality of life scale | For all 24 CTD patients: At V1 (Day1/Day2) For 9 out of 24 CTD patients: Repeated at V3 (Day30) and V7 (Day90).
  Quality of life scale (PedsQL 4.0 for children or San Martin scale if the patient is older than 18)
Cognitive assessments : Leiter 3 scale | For the 24 CTD patients: at V1 (Day1/Day2), For 9 out of 24 CTD patients: repeated at V7 (Day90). Controls: Cognitive assessment at V1(Day 1)
  Leiter 3 scale (4 cognitive sub-tests to be able to compute the non-verbal IQ and 2 non-verbal memory sub-tests) or Bayley 4 if Leiter 3 is not possible
Cognitive assessments : CPM-BF | For the 24 CTD patients: at V1 (Day1/Day2), For 9 out of 24 CTD patients: repeated at V7 (Day90). Controls: Cognitive assessment at V1(Day 1)
  CPM-BF : Raven's coloured Progressive Matrices
Cognitive assessments : reasoning task | For the 24 CTD patients: at V1 (Day1/Day2), For 9 out of 24 CTD patients: repeated at V2 (Day15), V3 (Day30), V4 (Day45), V5 (Day60), V6 (Day75) and V7 (Day90). Controls: Cognitive assessment at V1(Day 1)
  Simple reasoning task on tablet (match-to-sample task)
Cognitive assessments : Implicit rules learning | For the 24 CTD patients: at V1 (Day1/Day2), For 9 out of 24 CTD patients: repeated at V2 (Day15), V3 (Day30), V4 (Day45), V5 (Day60), V6 (Day75) and V7 (Day90). Controls: Cognitive assessment at V1(Day 1)
  Implicit rules learning (modified Brixton),
Cognitive assessments : WPPSI-IV | For the 24 CTD patients: at V1 (Day1/Day2), For 9 out of 24 CTD patients: repeated at V3 (Day30) and V7 (Day90). Controls: Cognitive assessment at V1(Day 1)
  4 sub-tests from the WPPSI-IV ("zoo location" to assess spatial memory, "block design" to assess visuo-constructive abilities, "bug search" , "cancellation"),
Cognitive assessments : Attention assessment | For the 24 CTD patients: at V1 (Day1/Day2), For 9 out of 24 CTD patients: repeated at V3 (Day30) and V7 (Day90). Controls: Cognitive assessment at V1(Day 1)
  Attention assessment (4 sub-tests from KITTAP: alert, go/no go, flexibility, divided attention),
Cognitive assessments : Elementary visuo-spatial perception | For the 24 CTD patients: at V1 (Day1/Day2), For 9 out of 24 CTD patients: repeated at V2 (Day15), V3 (Day30), V4 (Day45), V5 (Day60), V6 (Day75) and V7 (Day90). Controls: Cognitive assessment at V1(Day 1)
  Elementary visuo-spatial perception (on tablets)
Language assessments : EXALANG 3-6 | For all 24 CTD patients: performed at V1 (Day1/Day2). For 9 out of 24 CTD patients: repeated at V3 (Day30), and V7 (Day90). Controls: Language assessment at V1(Day 1)
  EXALANG 3-6 - Computerized battery for the evaluation of oral and written language : 10 sub-tests testing for expressive and receptive language assessments
Language assessments : vocabulary | For all 24 CTD patients: performed at V1 (Day1/Day2). For 9 out of 24 CTD patients: repeated at V3 (Day30), and V7 (Day90). Controls: Language assessment at V1(Day 1)
  PPVT-5 : Peabody Picture Vocabulary Test Fifth Edition = receptive vocabulary, EVT-3 : Expressive Vocabulary Test third edition,
Language assessments : Automatic language analysis | For all 24 CTD patients: performed at V1 (Day1/Day2). For 9 out of 24 CTD patients: repeated at V3 (Day30), and V7 (Day90). Controls: Language assessment at V1(Day 1)
  Automatic language analysis (during a 10 minutes interaction, play).
Motor assessments : Kinematic task | CTD patients : performed at V1 (Day1/Day2). Controls: Motor assessment at V1 (Day 1)
  Kinematic task (specifically designed)
Motor assessments : Purdue-Pegboard test | CTD patients : performed at V1 (Day1/Day2), V3(Day30), and V7 (Day90). Controls: Motor assessment at V1 (Day 1)
  Purdue-Pegboard test
Motor assessments : Renzi test | CTD patients : performed at V1 (Day1/Day2), V3(Day30), and V7 (Day90). Controls: Motor assessment at V1 (Day 1)
  Renzi test
Social assessments : Eye-tracking | CTD patients : performed at V1 (Day1/Day2), V3 (Day30) and V7 (Day90). Controls : Social assessment at V1(Day1)
  Eye-tracking analysis of social visual scenes and social preference index (movies)
Social assessments : Theory of mind assessment | CTD patients : performed at V1 (Day1/Day2). Controls : Social assessment at V1(Day1)
  Theory of mind assessment
Social assessments : ADOS scale (Autism Diagnostic Observation Scale) | CTD patients : performed at V1 (Day1/Day2). Controls : Social assessment at V1(Day1)
  ADOS scale (Autism Spectrum Disorder)
Social assessments : Sensitivity to inequality | CTD patients : performed at V1 (Day1/Day2). Controls : Social assessment at V1(Day1)
  Sensitivity to inequality
Social assessments : Pro-social behaviors (help of the psychologist) | CTD patients : performed at V1 (Day1/Day2). Controls : Social assessment at V1(Day1)
  Pro-social behaviors (help of the psychologist)

SECONDARY OUTCOMES:
Neuroimaging (MRI) | V1 (Day1/Day2)
  The MRI will be performed to describe structural and functional neuroanatomical profile of CTD patient in comparison to chronological age-matched controls and variability in creatine peak assessment using MR spectroscopy
Cardiac assessments : Electrocardiogram | CTD patients: V1 (Day1/Day2)
  Electrocardiogram (ECG) will be performed to describe CTD patients cardiac profile (especially the risk of increased QTC and/or cardiac echography abnormality)
Cardiac assessments : Ultrasound | CTD patients: V1 (Day1/Day2)
  Cardiac Ultrasound will be performed to describe CTD patients cardiac profile (especially the risk of increased QTC and/or cardiac echography abnormality)
Biological collection : Blood sample | CTD patients: V1 (Day1/Day2)
  Blood sample (plasma and peripheral blood mononuclear cells)
Biological collection : Urine sample | CTD patients: V1 (Day1/Day2)
  Urine sample will be collected to create a collection of biological samples associated with clinical and genomic data from CTD patients. In the future this will be usefull for research labs to investigate new biomarkers (not identified yet) or to test for the efficiency of new therapeutic approaches in vitro (on cultivated fibroblasts or after the development of iPS cells or organoïds) in this rare disease.
Biological collection : Superficial skin biopsy | CTD patients: V1 (Day1/Day2)
  Superficial skin biopsy will be performed to get cultivated fibroblasts to create a collection of biological samples associated with clinical and genomic data from CTD patients. In the future this will be usefull for research labs to investigate new biomarkers (not identified yet) or to test for the efficiency of new therapeutic approaches in vitro (on cultivated fibroblasts or after the development of iPS cells or organoïds) in this rare disease.
Biological collection : biological profile of DTC patients compared to sex- and chronological age-matched controls | Up to 12 months
  To describe the biological profile of DTC patients compared to sex- and chronological age-matched controls.
  Biological profile will be performed for CTD patients and the sex- and chronological age- matched controls who agreed on participating to the biological collection.

CONTACTS AND LOCATIONS:
Locations (1):
- Woman, mother and child hospital, Hospices Civils de Lyon, Bron, France

IPD SHARING:
Plan to Share IPD: No